CLINICAL TRIAL: NCT06357611
Title: Effect of the Muscular Energy Technique With the 4th Ventricle Technique on the Range of Motion of the Hamstring Muscles in Female Basketball Players: RCT
Brief Title: Combination of Two Osteopathic Techniques for the Hamstring's Stretching Capacity in Basketball Female Players
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Natália Maria Oliveira Campelo (Other)
Responsible Party: Sponsor-Investigator, Natália Maria Oliveira Campelo, Profesor, Escola Superior de Tecnologia da Saúde do Porto
Organization: Escola Superior de Tecnologia da Saúde do Porto (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: OST1_015
Record Dates: First submitted 2024-04-05; First posted 2024-04-10 (Actual); Last update posted 2024-04-30 (Actual); Status verified 2024-04

CONDITIONS: Healthy
Keywords: Fourth ventricle technique; Muscle energy technique; Range of motion; Hamstring Muscles

STUDY DESIGN:
Intervention Model Description: In order to allocate each participant to an intervention group, each voluntary participation questionnaire was assigned a number. Subsequently, all the numbers of the participants in the sample were randomly distributed among the 3 groups by the principal investigator.
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control Group (Placebo Comparator): After completing an individual questionnaire and giving informed consent, a placebo technique was performed, consisting only of contact in the area of the participant's shoulders.
  Interventions: Other: Simulated technique
- Experimental group MET (Experimental): After completing an individual questionnaire and giving informed consent, the muscle energy technique was performed on the dominant hamstring muscle.
  Interventions: Other: Muscle energy technique
- Experimental group CV-4 and MET (Experimental): After completing an individual questionnaire and giving informed consent, the 4th ventricle technique (CV-4) was performed, followed by the muscle energy technique on the dominant hamstring muscle.
  Interventions: Other: 4th ventricle technique and muscular energy technique

INTERVENTIONS:
Other: Simulated technique — The participant was in a supine position, with her upper limbs at her sides and her neck in a neutral position.
  The researcher sat in a cephalic position, making contact with the participant's shoulders, without any movement, until 5 minutes had elapsed.
  Arms: Control Group
Other: Muscle energy technique — The participant was in a supine position, with her upper limbs alongside her body and her neck in a neutral position.
  The researcher adopted a position homolateral to the dominant limb, contacting the lower limb with the caudal hand in the region of the malleoli. He then helped the participant to perform the movement, which consisted of flexing the hip and extending the knee passively until the motor barrier was reached, and instructed her to perform an isometric contraction of the hamstrings. She was asked to perform three 7-second contractions with a 2 to 3-second interval, using approximately 20% of her maximum strength, gaining a new motor barrier between each set, for a total of three sets.
  Arms: Experimental group MET
Other: 4th ventricle technique and muscular energy technique — The participant was in a supine position, with her upper limbs alongside her body and her neck in a neutral position.
  For CV-4, the researcher contacted the squamous portion of the occiput laterally, bringing it close to the posterior convexity of the occiput, bringing the skull into extension, changing the compression movement with decompression, until 3 minutes had elapsed.
  For the MET, the researcher adopted a position homolateral to the dominant limb, contacting the lower limb with the caudal hand in the region of the malleoli. She then helped the participant to perform the movement, which consisted of flexing the hip and extending the knee passively to the motor barrier, having been instructed to perform an isometric contraction of the hamstring. A total of 3 7-second contractions with a 2-3 second interval were requested, using approximately 20% of her maximum strength, and with a new motor barrier being gained between each series, for a total of 3 series.
  Arms: Experimental group CV-4 and MET

SUMMARY:
It is known that there are studies that prove the effectiveness of muscle energy techniques and the fourth ventricle technique separately, however, information is scarce regarding the combination of the two and their effectiveness in the population. The aim of this randomized controlled study is to compare the immediate effects of the techniques compared to the muscle energy technique alone in female basketball players.

DETAILED DESCRIPTION:
The muscular energy technique (MET) is a manual therapy technique that uses isometric contractions with the aim of increasing the extensibility of the muscle group, as well as promoting lymphatic and venous circulation. The fourth ventricle technique (CV-four) plays an amplifying role in the movement of tissues and fluids, restoring the flexibility of the autonomous response. For the MET, the researcher adopted a position homolateral to the dominant limb, contacting the lower limb with the caudal hand in the region of the malleoli. He then helped the participant to perform the movement, which consisted of flexion of the hip and extension of the knee passively until the motor barrier was reached, after which she was instructed to perform an isometric contraction of the hamstring. A total of three contractions of seven seconds with an interval of two to three seconds were requested, using approximately twenty per cent of their maximum force, and gaining a new motor barrier between each series, for a total of three series. For the CV-four technique, the researcher adopted a seated position and laterally contacted the scaly portion of the occiput, bringing it closer to the posterior convexity of the occiput, bringing the skull into extension, changing the compression movement with decompression, until three minutes had elapsed. At all stages of the session, the participant was positioned in the supine position, with the upper limbs alongside the body and the neck in a neutral position. All the participants in the study underwent an initial and final assessment protocol to determine their range of motion (ROM).

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years old
* Female
* Playing federated basketball
* Signature of informed consent documents

Exclusion Criteria:

* Surgical intervention/trauma in the areas of activity (cervical-cranial and lower limb)
* Exposure to medicinal therapy
* Participants with hypertension
* Participants at risk of cerebral hemorrhage (e.g. aneurysm)

Ages: 18 Years to 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-09 (Estimated); Primary Completion 2024-12 (Estimated); Study Completion 2024-12 (Estimated)

PRIMARY OUTCOMES:
Altered range of motion of the hamstring muscles. | 10 minutes after intervention.
  The universal goniometer is a tool used to assess joint ROM.

CONTACTS AND LOCATIONS:
Overall Officials: Natália MO Campelo, PhD, Principal Investigator — Escola Superior de Saúde do Politecnico do Porto
Locations (1):
- Escola Superior de Saúde do Porto, Porto, Portugal

REFERENCES:
- [Background] Balasubramaniam, A., Gandhi V, M., Purushothaman, V. K. (2022). Myofascial Release Theraphy versus Muscle Energy Technique on Hamstring Flexibility in Physical Inactive students - A randomized controlled trial. Universal Journal of Public Health, 299-303.
- [Background] Barroso, G. C., & Thiele, E. S. (2011, Junho 28). Lesão Muscular nos Atletas.
- [Background] Bonorino, D. S. (2017). Efeitos da técnica CV-4 para o tratamento da enxaqueca.
- [Background] Chaitow, L. (2013). Muscle Energy Techniques.
- [Background] Chaitow, L. (2023). Muscle Energy Techniques (Fifth Edition ed.). Elsevier.
- [Background] DeLucia, R. (2016). Farmacologia Integrada: Uso Racional de Medicamentos.
- [Background] DeStefano, L. (2011). Principales of Manual Medicine. Wolters Kluwer.
- [Background] E. de Gray, L., & Seth, B. (2020). Drugs used to treat joint and muscle disease.
- [Background] Favareto, R. M. (2019). Influência da manipulação osteopática craniana, sobre o sistema nervoso autônomo mensurado pela neurometria funcional em pacientes com fibromialgia. Revista Científica de Neurometria, 5.
- [Background] Fryer, G., Fleischmann, M., & Vaughan, B. (2021). Use of muscle energy technique amongst a nationally representative sample of Australian Osteopaths. International Journal of Osteopathic Medicine, 5.
- [Background] Jakel A, von Hauenschild P. Therapeutic effects of cranial osteopathic manipulative medicine: a systematic review. J Am Osteopath Assoc. 2011 Dec;111(12):685-93. PMID 22182954
- [Background] Kang YH, Ha WB, Geum JH, Woo H, Han YH, Park SH, Lee JH. Effect of Muscle Energy Technique on Hamstring Flexibility: Systematic Review and Meta-Analysis. Healthcare (Basel). 2023 Apr 11;11(8):1089. doi: 10.3390/healthcare11081089. PMID 37107922
- [Background] Laurino, C., Murer, F., & Iglesias, R. (2018, Julho 19). Tratamento cirurgico das lesões dos músculos isquiotibiais da coxa.
- [Background] Liem, T. (2004). Cranial Osteopathy: principles and practice. Elsevier.
- [Background] Nicholas, A. N. (2016). Atlas of Osteopathic Techniques (3 ed.). Wolters Kluwer Editora.
- [Background] Parsons, J., & Marcer, N. (2008). Osteopathy: Models for Diagnosis, Treatment and Practice. Elsevier.
- [Background] Ricard, F., & Sallé, J.-L. (2010). Tratado de Osteopatía.
- [Background] Smith M, Fryer G. A comparison of two muscle energy techniques for increasing flexibility of the hamstring muscle group. J Bodyw Mov Ther. 2008 Oct;12(4):312-7. doi: 10.1016/j.jbmt.2008.06.011. Epub 2008 Aug 6. PMID 19083689
- [Background] Upledger, J. E., & Vredevoogd, J. D. (1983). Craniosacral therapy (Vol. 236). Seattle: Eastland press.